CLINICAL TRIAL: NCT02354781
Title: Phase I/II Clinical Intramuscular Gene Transfer of rAAV1.CMV.huFollistatin344 Trial to Patients With Duchenne Muscular Dystrophy
Brief Title: Clinical Intramuscular Gene Transfer of rAAV1.CMV.huFollistatin344 Trial to Patients With Duchenne Muscular Dystrophy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jerry R. Mendell (Other)
Collaborators: Duchenne Alliance (Other); Milo Therapeutics (Industry)
Responsible Party: Sponsor-Investigator, Jerry R. Mendell, Center Director for Gene Therapy, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 14-00630
Record Dates: First submitted 2015-01-26; First posted 2015-02-03 (Estimated); Results first posted 2020-04-15 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-09

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: DMD; muscular dystrophy; Follistatin
MeSH Terms: conditions — Muscular Dystrophy, Duchenne; Muscular Dystrophies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Experimental (Experimental): The vector will be delivered to both limbs via multiple, direct intramuscular injections of rAAV1.CMV.huFollistin344; the number of injections per muscle will depend on the size of the patient. A total dose of 2.4E12 vg/kg (1.2E12vg/kg/limb) will be delivered to the lower limbs of 6 DMD subjects
  Interventions: Biological: rAAV1.CMV.huFollistin344

INTERVENTIONS:
Biological: rAAV1.CMV.huFollistin344 — Six DMD patients will receive rAAV1.CMV.huFollistatin344 to both limbs by multiple injections to gluteal muscles, quadriceps and tibialis anterior muscles.

SUMMARY:
The proposed clinical trial is an outgrowth of the safety record and functional improvement seen in the BMD follistatin gene therapy trial. In this study the investigators propose to inject AAV1.CMV.huFS344 at a total dose of 2.4E12 vg/kg to six DMD patients. This dose will be divided between gluteal muscles, quadriceps and tibialis anterior. This is a wider distribution of vector than given to BMD patients, who overall improved the distance walked on the 6MWT without adverse events related to viral transduction into a single muscle.

DETAILED DESCRIPTION:
The primary objective of this study is safety and endpoints will include hematology, serum chemistry, urinalysis, immunologic response to rAAV1 and follistatin, and reported history and observations of symptoms. Efficacy measures will be used as secondary outcomes and include the distance walked on the 6MWT, functional tests by PT, life quality questionnaire, MRI, EIM, and muscle biopsy. Subject will have follow up visits on days 7, 14, 30, 45, 60, 90, 180 and 9,12, 18 and 24 months post-gene transfer.

ELIGIBILITY:
Inclusion Criteria:

* Age 7 or older
* Confirmed DMD gene mutations
* Impaired muscle function based on clinical evidence including difficulty climbing stairs, getting from the floor (Gowers' sign), and weakness of individual muscles of extremities
* Males of any ethnic group will be eligible
* Ability to cooperate with study procedures including muscle testing.
* Willingness of sexually active subjects with reproductive capacity to practice reliable method of contraception
* Subjects must be on stable dose of prednisone for three months at time of enrollment or be started on oral dose of daily prednisone regimen for 30 days prior to gene transfer. Study participants will continue prednisone post gene transfer unless there is adverse event that warrants prednisone taper or withdrawal.

Exclusion Criteria:

* Active viral infection based on clinical observations.
* The presence of a DMD gene mutation without weakness or loss of function
* Symptoms or signs of cardiomyopathy, including:
* Dyspnea on exertion, pedal edema, shortness of breath upon lying flat, or rales at the base of the lungs
* Echocardiogram with ejection fraction below 40%
* Serological evidence of HIV infection, or Hepatitis A, B or C infection
* Diagnosis of (or ongoing treatment for) an autoimmune disease
* Concomitant illness or requirement for chronic drug treatment that in the opinion of the PI creates unnecessary risks for gene transfer
* Subjects with rAAV1 binding antibody titers > 1:50 as determined by ELISA immunoassay
* Abnormal laboratory values for liver, kidney, CBC, in the clinically significant range, based upon normal values in the Nationwide Children's Hospital Laboratory

Min Age: 7 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2015-01; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jerry R Mendell, MD, Principal Investigator — Director, Center for Gene Therapy, Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

REFERENCES:
- [Background] Mendell JR, Sahenk Z, Malik V, Gomez AM, Flanigan KM, Lowes LP, Alfano LN, Berry K, Meadows E, Lewis S, Braun L, Shontz K, Rouhana M, Clark KR, Rosales XQ, Al-Zaidy S, Govoni A, Rodino-Klapac LR, Hogan MJ, Kaspar BK. A phase 1/2a follistatin gene therapy trial for becker muscular dystrophy. Mol Ther. 2015 Jan;23(1):192-201. doi: 10.1038/mt.2014.200. Epub 2014 Oct 17. PMID 25322757
- [Background] Kota J, Handy CR, Haidet AM, Montgomery CL, Eagle A, Rodino-Klapac LR, Tucker D, Shilling CJ, Therlfall WR, Walker CM, Weisbrode SE, Janssen PM, Clark KR, Sahenk Z, Mendell JR, Kaspar BK. Follistatin gene delivery enhances muscle growth and strength in nonhuman primates. Sci Transl Med. 2009 Nov 11;1(6):6ra15. doi: 10.1126/scitranslmed.3000112. PMID 20368179
- [Background] Rodino-Klapac LR, Haidet AM, Kota J, Handy C, Kaspar BK, Mendell JR. Inhibition of myostatin with emphasis on follistatin as a therapy for muscle disease. Muscle Nerve. 2009 Mar;39(3):283-96. doi: 10.1002/mus.21244. PMID 19208403
- [Background] Miller TM, Kim SH, Yamanaka K, Hester M, Umapathi P, Arnson H, Rizo L, Mendell JR, Gage FH, Cleveland DW, Kaspar BK. Gene transfer demonstrates that muscle is not a primary target for non-cell-autonomous toxicity in familial amyotrophic lateral sclerosis. Proc Natl Acad Sci U S A. 2006 Dec 19;103(51):19546-51. doi: 10.1073/pnas.0609411103. Epub 2006 Dec 12. PMID 17164329
- [Derived] Bian X, Snow ZK, Zinn CJ, Gowan CC, Conley SM, Bratulin AL, Elhusseiny KM, Miller J, Tchkonia T, Kirkland JL, Lerman LO, Hickson LJ. Activin A Antagonism with Follistatin Reduces Kidney Fibrosis, Injury, and Cellular Senescence-Associated Inflammation in Murine Diabetic Kidney Disease. Kidney360. 2025 Mar 28;6(8):1278-1291. doi: 10.34067/KID.0000000776. PMID 40152935
- See also: Click here for Center for Gene Therapy, The Research Institute at Nationwide Children's Hospital — http://www.nationwidechildrens.org/center-for-gene-therapy

RESULTS

PARTICIPANT FLOW:
Groups:
- 2.4E12 vg/kg CMV.huFollistatin344: Participants enrolled will receive a single dose of 2.4E12 vg/kg (1.2E12vg/kg/limb) of rAAV1.CMV.huFollistatin344 delivered to the lower limbs
Period: Overall Study
Arm/Group | 2.4E12 vg/kg CMV.huFollistatin344
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The Safety Population included all subjects who received one dose of 2.4E12 vg/kg (1.2E12vg/kg/limb) of rAAV1.CMV.huFollistatin344. The Safety Population is the primary analysis population for safety assessments
Groups:
- Dose Group 1: Participants enrolled will receive a single dose of 2.4E12 vg/kg (1.2E12vg/kg/limb) of rAAV1.CMV.huFollistatin344 delivered to the lower limbs
Arm/Group | Dose Group 1
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Dose Limiting Toxicity (DLT) Adverse Events as Assessed by 21 CFR 312.32.
Description: Dose limiting toxicity (DLT) is defined as any adverse event that is possibly, probably, or definitely related to the study agent. This would include any grade 3 according to the classification given above. Study enrollment will be halted by the investigators when any subject experiences a Grade 3, or higher adverse event toxicity that is possibly, probably, or definitely related to the study drug. Only those adverse events requiring treatment will qualify as DLT.
  The classification for adverse events to be used is the following:
  1. Mild adverse event; did not require treatment
  2. Moderate adverse event; resolved with treatment
  3. Severe adverse event; inability to carry on normal activities; required professional medical attention
  4. Life-threatening or permanently disabling adverse event
  5. Fatal adverse event In this grading system, "severe" is not equivalent to seriousness.
Time Frame: DLT Adverse events will be recorded from the date of dosing and through the time of the subject's last study visit. Serious adverse events will be recorded from the date of dosing and for up to 2 years after gene therapy administration.
Population: Safety Population: All subjects who receive a single total dose of 2.4E12 vg/kg (1.2E12vg/kg/limb) of rAAV1.CMV.huFollistatin344.
Measure: Number; unit: Number of Events
Groups:
- 2.4E12 vg/kg CMV.huFollistatin344: Participants enrolled who receive a total dose of 2.4E12 vg/kg (1.2E12vg/kg/limb) of rAAV1.CMV.huFollistatin344.
Arm/Group | 2.4E12 vg/kg CMV.huFollistatin344
Number analyzed (Participants) | 3
Number of Events | 0

2. Secondary Outcome: Muscle Function Measured by Six-minute Walk Test (6MWT)
Description: Number of subjects with increased distance walked in meters on the Six Minute Walk Test. The participant was asked to walk a set course of 25 meters for 6 minutes (timed) and the distance walked in meters was recorded. Increases from baseline in 6MWT distance are indicative of improvement and decreases from baseline indicate worsening.
Time Frame: 2 years
Population: Participants enrolled will receive a single dose of 2.4E12 vg/kg (1.2E12vg/kg/limb) of rAAV1.CMV.huFollistatin344 delivered to the lower limbs
Measure: Count of Participants; unit: Participants
Groups:
- 2.4E12 vg/kg CMV.huFollistatin344: Participants enrolled will receive a total dose of 2.4E12 vg/kg (1.2E12vg/kg/limb) of rAAV1.CMV.huFollistatin344 delivered to the lower limbs
Arm/Group | 2.4E12 vg/kg CMV.huFollistatin344
Number analyzed (Participants) | 3
Participants | 0

3. Secondary Outcome: Expression of Viral DNA (qPCR), and Follistatin Transgene in Muscle Tissue
Description: Muscle biopsies on quadriceps muscles a muscle biopsy on one leg at baseline screening visit and the post gene transfer biopsy on the opposite leg at day 180. Muscle tissue obtained at biopsy will also be assessed for viral DNA (qPCR), and follistatin transgene expression.
  Measured in CMV.FS344 Gene Copy Number in Genomic DNA (Copies/ug DNA)
Time Frame: 180.days
Population: All muscle biopsies were canceled per PI discretion due to the disease progression of each participant.
Arm/Group | 2.4E12 vg/kg CMV.huFollistatin344
Number analyzed (Participants) | 0

4. Secondary Outcome: Improvement of Muscle Function as Measured by North Star Ambulatory Assessment (NSAA)
Description: Overall Improvement in North Star Ambulatory Assessment
  The activities are graded as follows:
  2 - "Normal" - no obvious modification of activity
  1 - Modified method but achieves goal independent of physical assistance from another 0 - Unable to achieve independently This scale is ordinal with 34 as the maximum score indicating fully-independent function.
Time Frame: 2 years
Population: Participants enrolled who receive a single dose of 2.4E12 vg/kg (1.2E12vg/kg/limb) of rAAV1.CMV.huFollistatin344.
Measure: Count of Participants; unit: Participants
Arm/Group | 2.4E12 vg/kg CMV.huFollistatin344
Number analyzed (Participants) | 3
Participants | 1

ADVERSE EVENTS:
Time Frame: Adverse events will be recorded from the date of informed consent and for up to 2 years after gene therapy administration, the subject's last study visit. Serious adverse events will be recorded from the date of informed consent and for up to 2 years after gene therapy administration, the subject's last study visit.
Groups:
- 2.4E12 vg/kg (1.2E12vg/kg/Limb) of rAAV1.CMV.huFollistatin344: Participants enrolled will receive a total dose of 2.4E12 vg/kg (1.2E12vg/kg/limb) of rAAV1.CMV.huFollistatin344 delivered to the lower limbs
Arm/Group | 2.4E12 vg/kg (1.2E12vg/kg/Limb) of rAAV1.CMV.huFollistatin344
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 1/3
Other Adverse Events (participants affected / at risk) | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2.4E12 vg/kg (1.2E12vg/kg/Limb) of rAAV1.CMV.huFollistatin344 (N=3)
Head Injury From Fall (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2.4E12 vg/kg (1.2E12vg/kg/Limb) of rAAV1.CMV.huFollistatin344 (N=3)
Pain (Injury, poisoning and procedural complications) | 3 (5)
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Abrasion (Skin and subcutaneous tissue disorders) | 1 (2)
Anxiety (Psychiatric disorders) | 1 (2)
Behavioral Changes/Agitation (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Bruising (Skin and subcutaneous tissue disorders) | 2 (3)
GERD (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Stye (Eye disorders) | 1 (1)
Increased Muscle Weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Compression Fracture (Injury, poisoning and procedural complications) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Influenza (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-01-16): https://cdn.clinicaltrials.gov/large-docs/81/NCT02354781/Prot_SAP_000.pdf